CLINICAL TRIAL: NCT06449898
Title: Validity and Reliability of the Turkish Version of the Ottawa Sitting Scale in Hemodialysis Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Hanifi Kaya, Pilot Project Manager Lecturer Doctor., Kirsehir Ahi Evran Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023/04
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The sample size was determined based on the recommendations for validation studies, which suggest a minimum of 5 to 10 participants per item on the scale being validated. Given that the OSS comprises 12 items, a minimum of 60 participants was deemed necessary. However, to account for potential dropouts and to enhance the robustness of the findings, 130 participants were recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hemodialysis group (Other): Undergoing hemodialysis treatment for at least 6 months.
  Interventions: Other: hemodialysis group

INTERVENTIONS:
Other: hemodialysis group — Data were collected from patients undergoing treatment at a hemodialysis center in Kırşehir. Participants were informed about the study objectives and provided written consent. Data collection took approximately 20-30 minutes per participant and included a face-to-face interview where socio-demographic and clinical information was recorded.

SUMMARY:
Background:

Prolonged sitting behavior, characterized by minimal energy expenditure, poses significant health risks, especially for chronic kidney disease (CKD) patients undergoing hemodialysis. This sedentary behavior can lead to various health complications and a reduced quality of life (QOL).

Objectives:

This study aims to evaluate the validity and reliability of the Turkish adaptation of the Ottawa Sitting Scale (OSS) in assessing sitting behavior among CKD patients.

Methods:

A total of 130 CKD patients undergoing hemodialysis participated in this cross-sectional study conducted in XXX province between January 2023 and September 2023. The OSS, along with the Physical Activity Scale (FAS), Sitting Behavior Assessment (SBA), and Quality of Life Scale (QOL), was administered. Data analysis involved assessing the internal consistency, factor structure, and concurrent validity of the OSS.

DETAILED DESCRIPTION:
Prolonged sitting behavior, characterized by minimal energy expenditure, poses significant health risks, especially for chronic kidney disease (CKD) patients undergoing hemodialysis. This sedentary behavior can lead to various health complications and a reduced quality of life.This study aims to evaluate the validity and reliability of the Turkish adaptation of the Ottawa Sitting Scale (OSS) in assessing sitting behavior among CKD patients. A total of 130 CKD patients undergoing hemodialysis participated in this cross-sectional study conducted in XXX province between January 2023 and September 2023. The OSS, along with the Physical Activity Scale (FAS), Sitting Behavior Assessment (SBA), and Quality of Life Scale (QOL), was administered. Data analysis involved assessing the internal consistency, factor structure, and concurrent validity of the OSS.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of CKD undergoing hemodialysis treatment for at least 6 months no abnormalities in cooperation or communication, and willingness to participate in the study.

Exclusion Criteria:

* Inability to comprehend instructions
* Presence of any other disease that may affect sitting
* Experiencing acute or chronic musculoskeletal injuries, pain, inflammation or deformities, and refusal to participate in the study.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Ottawa Sitting Scale (OSS): | 24 weeks
  The OSS is a 6-item scale designed to assess sitting balance. Each item is performed with feet supported and unsupported, resulting in a total of 12 items. A 4-point Likert-type response scale was used for each item. The total score ranges from 0 to 48, with higher scores indicating better sitting behavior. The cross-cultural adaptation of the OSS followed the guidelines by Beaton et al. (2000), involving forward and backward translations, synthesis, expert committee review, and pre-testing on 30 elderly adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Hanifi KAYA, Kırşehir, Turkey (Türkiye)